CLINICAL TRIAL: NCT02242071
Title: The Effect of Autologous Bone Marrow Mononuclear Cell Transplantation on Motor Neuron Disease/Amyotrophic Lateral Sclerosis
Brief Title: Cell Therapy for Motor Neuron Disease/Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-10
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Autologous Mononuclear Cell therapy; Stem cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental): bone marrow mononuclear cell transplantation
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — intrathecal autologous bone marrow mononuclear cell transplantation

SUMMARY:
The effect of autologous bone marrow mononuclear cells on Motor Neuron Disease/Amyotrophic Lateral Sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of definite Motor Neuron Disease/amyotrophic lateral sclerosis.
* Age 18-80 years

Exclusion Criteria:

* HIV/HBV/HCV
* Malignancies
* Bleeding tendencies
* Pneumonia
* Renal failure
* Severe liver dysfunction
* Severe anemia [hb < 8]
* Any bone marrow disorder
* Space occupying lesion in brain
* Pregnancy and lactation
* Other acute medical conditions/infections such as respiratory infection and pyrexia
* left ventricular ejection fraction < 25%
* Patient on artificial ventilatory support

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2015-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional rating scale-revised | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No